CLINICAL TRIAL: NCT03716076
Title: The Effect of Carbetocin Dose on Dispersion of Myocardial Repolarization in Healthy Parturients Scheduled for Elective Cesarean Delivery Under Spinal Anesthesia
Brief Title: Carbetocin on Myocardial Repolarization Dynamics in Obstetrics Study
Acronym: CaRDIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: H18-02232
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrythmias
Keywords: Carbetocin; Myocardial repolarization
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant receives 50 mcg of carbetocin post-delivery. (Experimental): Participant receives 50 mcg of carbetocin post-delivery.
  Interventions: Drug: Carbetocin
- Participant receives 100 mcg of carbetocin post-delivery. (Experimental): Participant receives 100 mcg of carbetocin post-delivery.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — 50 mcg or 100 mcg bolus of carbetocin

SUMMARY:
Relationship between carbetocin dose on transmural dispersion of repolarization (TDR).

DETAILED DESCRIPTION:
Carbetocin is a uterotonic used to prevent postpartum hemorrhage. Although it has been proven to be completely safe, little is known about its effects on the electrical activity of the heart. The investigators aim to determine its effect on myocardial repolarization dynamics

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients ≥ 36 weeks gestation, for elective Cesarean delivery under neuraxial anesthesia
* American Society of Anesthesiologists (ASA) class 2
* Patients ≥ 19 years of age

Exclusion Criteria:

* Long QT syndrome
* Cardiac disease or rhythm abnormalities
* Family history of long QT syndrome or abnormal cardiac conduction
* Currently taking medication that is known to prolong the QT interval
* Women who are high risk for uterine atony as outlined in SOGC
* Known allergic reaction or hypersensitivity to Carbetocin or any other oxytocin homologue
* Patients who are unable to give informed consent because of a language barrier as the study team only speaks English and will be unable to complete consent process and study procedure appropriately.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD MMSc, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clunies-Ross N, Roston TM, Taylor J, Whyte S, Albert A, Gorges M, Chau A. The Effect of Carbetocin Dose on Transmural Dispersion of Myocardial Repolarization in Healthy Parturients Scheduled for Elective Cesarean Delivery Under Spinal Anesthesia: A Prospective, Randomized Clinical Trial. Anesth Analg. 2021 Feb 1;132(2):485-492. doi: 10.1213/ANE.0000000000004712. PMID 32149759

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Started | 25 | 25
Completed | 22 | 19
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery. | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (4.3) | 35.7 (2.8) | 35 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 19 | 41
Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] | 89.7 (10.4) | 88.5 (8.3) | 89.2 (9.4)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 83.0 (8.6) | 81.8 (9.0) | 82.0 (8.7)
Gravida [Median (Inter-Quartile Range); unit: pregnancies] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Parity of 0 [Number; unit: participants] | 7 | 5 | 12
Gestational Age [Mean (Standard Deviation); unit: weeks] | 38.9 (0.8) | 39.2 (0.5) | 39.0 (0.7)
Parity greater than 0 [Number; unit: participants] | 15 | 14 | 29
Baseline QTc [Mean (Standard Deviation); unit: milliseconds] — Baseline Bazett-corrected Q-T interval
  milliseconds | 413.7 (11.0) | 409.0 (15.8) | 411.6 (13.5)
Baseline Tp-e [Mean (Standard Deviation); unit: milliseconds] — Time between peak and end of T-wave
  milliseconds | 67.5 (8.2) | 69.6 (5.7) | 68.5 (7.1)
Weight [Mean (Standard Deviation); unit: Kilograms] | 74.9 (13.2) | 75.1 (10.7) | 75.0 (12.0)
Phenylephrine Dose [Mean (Standard Deviation); unit: micrograms] | 1459.0 (426.1) | 1538.1 (479.2) | 1495.6 (500.2)

OUTCOME MEASURES:

1. Primary Outcome: Tp-e
Description: Time interval between peak and end of T-wave (Tp-e)
Time Frame: 5 minutes post-carbetocin administration
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
milliseconds | 69.5 (7.7) | 74.7 (4.7)
Statistical Analysis 1: Comparison: Participant Receives 50 mcg of Carbetocin Post-delivery. vs Participant Receives 100 mcg of Carbetocin Post-delivery; Test type: Other — mixed-effects linear regression; To compare time values to baseline, post-hoc Tukey's test was applied

2. Secondary Outcome: Arrhythmia
Description: Occurrence of Atrial or Ventricular Arrhythmias
Time Frame: perioperatively, typically ranging 30 minutes-1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
Participants | 0 | 0

3. Secondary Outcome: QTc at 5 Min
Description: Bazette corrected Q-T interval
Time Frame: 5 min post-carbetocin administration
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
milliseconds | 435.1 (18.3) | 434.2 (18.8)

4. Secondary Outcome: QTc 10 Min
Description: Bazette corrected Q-T interval (QTc)
Time Frame: 10 minutes post-carbetocin administration
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
milliseconds | 431.6 (18.2) | 431.9 (15.4)

5. Secondary Outcome: QTc 5 Min Spinal
Description: Bazette corrected Q-T interval change after spinal anesthesia
Time Frame: 5 min post-administration of spinal anesthesia
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
milliseconds | 409.4 (19.2) | 413.6 (17.4)

6. Secondary Outcome: Tp-e 5 Min Post-spinal
Description: Time between peak and end of T-wave,
Time Frame: 5 minutes after administration of spinal anesthesia
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
milliseconds | 69.5 (8.6) | 70.9 (6.5)

7. Secondary Outcome: Tp-e at 10 Min
Description: Time between peak and end of T-wave
Time Frame: 10 minutes post-carbetocin administration
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
Number analyzed (Participants) | 22 | 19
milliseconds | 69.4 (8.2) | 71.8 (5.5)

ADVERSE EVENTS:
Time Frame: 2 days, which is the typical time spent in hospital for monitoring after cesarean sections
Description: Participants are screened for a history of intolerance to oxytocin, which puts them at low risk of intolerance/mortality or serious adverse reaction to carbetocin.
  Patients are monitored for minor adverse events, such as arrhythmia, which are potential side effects of carbetocin dosing.
Arm/Group | Participant Receives 50 mcg of Carbetocin Post-delivery. | Participant Receives 100 mcg of Carbetocin Post-delivery.
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
No data exists that stratifies risk by measuring absolute Tp-e change We excluded patients with low repolarization reserves, or a resistance to oxytocin. We also excluded emergent C-sections, combined spinal/epidurals, and General Anesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT03716076/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT03716076/SAP_001.pdf